CLINICAL TRIAL: NCT01755182
Title: Randomized Phase 3 Trial Evaluating the Efficacy of Locoregional Treatment With Transarterial Embolization (TAE) for Liver Metastases, in Combination With Pharmacotherapy, in Patients With Neuroendocrine Tumor and Inoperable Liver Metastasis.
Brief Title: Systemic Therapy With or Without Upfront Transarterial Embolization for Inoperable Liver Metastasis of Neuroendocrine Tumors
Acronym: LOTUS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: difficulty enrollment, no patients received treatment
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: Federico II University (Other); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOTUS; 2011-006097-76 (EudraCT Number)
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Neuroendocrine Tumors
Keywords: locoregional treatment; liver metastases; transarterial embolization; upfront treatment; inoperable; octreotide; gastroenteropancreatic (GEP)primary; pulmonary primary; primary unknown origin; systemic therapy
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacologic therapy (Active Comparator): Patients in this arm receive systemic pharmacologic therapy alone
  Interventions: Drug: approved pharmacologic therapy
- TAE and pharmacologic therapy (Experimental): Patients in this arm receive systemic pharmacologic therapy and TAE
  Interventions: Drug: approved pharmacologic therapy; Procedure: TAE

INTERVENTIONS:
Drug: approved pharmacologic therapy
  Other Names: somatostatin analog or other medicine with proven efficacy
Procedure: TAE — after randomization, and after 3 months
  Other Names: transarterial embolization
  Arms: TAE and pharmacologic therapy

SUMMARY:
The purpose of this study is to verify if adding a locoregional treatment of liver metastasis (with trans-arterial embolization-TAE) to medical treatments of proven efficacy can prolong the progression free survival of patients affected by neuroendocrine tumors (NET) with inoperable liver metastases

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NET of gastroenteropancreatic (GEP), pulmonary or unknown primary site origin
* Unresectable liver metastases, according the judgment of surgeon, (the reasons for the opinion of surgeon should be made explicit)
* Hepatic involvement ≤50% volume of the organ
* Radiological evidence of hepatic lesions (contemporaneous progression or appearance of extrahepatic lesions are allowed if not critical sites) that require change or initiation of systemic pharmacotherapy
* Patients undergoing , previously treated , or never treated with systemic medical therapy are eligible
* Patients with or without carcinoid syndrome are eligible
* Well (G1) or medium (G2) differentiated histology (according to WHO 2010 classification)
* Ki67 ≤ 20% (G1-G2)
* Life expectancy > 6 months
* Age ≥ 18 and < 80 years

Exclusion Criteria:

* Previous loco-regional post-surgical treatment
* Poorly differentiated histology
* Severe concomitant morbidities such as: severe coagulopathy, severe liver failure (to be detailed), renal failure (creatinine > 2.0 mg/dl) and heart failure (NYHA 3-4 or unstable ischemic heart disease), contraindicating the interventional procedure or influencing the general prognosis (Investigator to provide details of exclusion)
* Extrahepatic metastasis in critical locations as: brain, spinal cord, lung with respiratory impairment, symptomatic vertebral lesions
* Patients with only extra-hepatic lesions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
progression free survival | two years

SECONDARY OUTCOMES:
overall survival | 3 years
number of objective responses | measured at 3 months and 6 months
changes in quality of life | up to 6 months
worst grade adverse event per patient | 6 months

OTHER OUTCOMES:
exploratory analysis of prognostic factors | 3 years
  clinical factors will be explored in relation to patient outcomes

CONTACTS AND LOCATIONS:
Overall Officials: A Colao, M.D., Principal Investigator — Federico II University; A Faggiano, M.D., Principal Investigator — Federico II University; R D'Angelo, M.D., Principal Investigator — NCI Naples; F Fiore, MD, Principal Investigator — NCI Naples; F Perrone, MD, Principal Investigator — NCI Naples; C Gallo, MD, Principal Investigator — University of Campania Luigi Vanvitelli; MC Piccirillo, MD, Principal Investigator — NCI Naples
Locations (12):
- Italy (12):
  - Albano Laziale Ospedale "Regina Apoltolorum", Albano Laziale
  - Università di Ferrara, Ferrara
  - Università di Genova, Genova
  - Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori, Milan
  - Ospedale San Raffaele, Milan
  - Istituto Nazionale dei Tumori, Napoli
  - Ospedale Cardarelli, Napoli
  - Presidio Monaldi - AORN Ospedale dei Colli, Napoli
  - Istituto Regina Elena, Roma
  - Azienda Ospedaliero-Universitaria S.M. della Misericordia di Udine, Udine
  - Università di Verona Policlinico GB Rossi, Verona